CLINICAL TRIAL: NCT00019097
Title: Phase II Study of Autologous Myeloma-Derived Immunoglobulin Idiotype Conjugated to Keyhole Limpet Hemocyanin Plus Sargramostim (GM-CSF) in Patients With Multiple Myeloma Undergoing Second Autologous Peripheral Blood Stem Cell Transplantation
Brief Title: Vaccine Therapy in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000064244; NCI-97-C-0033B; NCI-T94-0094N; CRB-9409; NCT00001562 (obsolete NCT alias)
Record Dates: First submitted 2007-03-01; First posted 2007-03-05 (Estimated); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Stage II Multiple Myeloma; Stage III Multiple Myeloma; Refractory Plasma Cell Neoplasm
Keywords: body system/site cancer; cancer; genetic condition; hematopoietic/lymphoid cancer; multiple myeloma; multiple myeloma and other plasma cell neoplasms; plasma cell neoplasm; refractory plasma cell neoplasm; stage II multiple myeloma; stage III multiple myeloma; stage, plasma cell neoplasm
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Neoplasms; Genetic Diseases, Inborn; Hematologic Neoplasms | interventions — FANG vaccine; keyhole-limpet hemocyanin; Melphalan; sargramostim

INTERVENTIONS:
Drug: autologous tumor cell vaccine
Drug: keyhole limpet hemocyanin
Drug: melphalan
Drug: sargramostim

SUMMARY:
RATIONALE: Vaccines made from a person's tumor cells may make the body build an immune response and kill their tumor cells. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy used to kill tumor cells.

PURPOSE: Phase II trial to study the effectiveness of peripheral stem cell transplantation plus vaccine therapy and chemotherapy in treating patients who have multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether autologous myeloma-derived immunoglobulin idiotype conjugated to keyhole limpet hemocyanin plus sargramostim (GM-CSF) can induce cellular and humoral immunity against the unique idiotype expressed on the surface of myeloma cells in patients with multiple myeloma undergoing second autologous peripheral blood stem cell transplantation.

II. Determine the clinical efficacy and safety of this regimen in these patients.

PROTOCOL OUTLINE: Within 6 months after the first autologous peripheral blood stem cell transplantation (APBSCT), patients receive melphalan IV over 30 minutes on day -2 and the second APBSCT on day 0. Sargramostim (GM-CSF) is administered subcutaneously (SC) beginning on day 1 and continuing until blood counts recover. Patients are also assigned to 1 of 3 vaccination groups.

Group 1: Patients receive autologous myeloma-derived immunoglobulin idiotype conjugated to keyhole limpet hemocyanin (Id-KLH) SC on day 1 and GM-CSF SC on days 1-4 of months 2, 3, and 5 after the second APBSCT for a total of 3 vaccinations.

Group 2: Patients receive Id-KLH SC on day 1 and GM-CSF SC on days 1-4 of months 2, 3, 4, 5, 6, and 8 after the second APBSCT for a total of 6 vaccinations.

Group 3: Patients receive Id-KLH SC on day 1 and GM-CSF SC on days 1-4 of weeks -8, -6, and -2 before and months 2, 3, and 5 after the second APBSCT for a total of 6 vaccinations.

Patients are followed within 3 months and then every 6 months.

PROJECTED ACCRUAL:

A maximum of 60 patients (20 per treatment group) will be accrued for this study within 3 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Immunoglobulin G or immunoglobulin A (IgA) multiple myeloma Low or intermediate risk disease based on the following criteria: Cytogenetics: no translocations, 11q, or -13/13q- Beta-2 microglobulin less than 2.5 mg/L before the first autologous peripheral blood stem cell transplantation (APBSCT) M-protein concentration in harvested plasma greater than 50% of total immunoglobulin of corresponding isotype (M-protein must be able to be purified by protein A- or anti-IgA-sepharose) Patients achieving partial or complete response after the first APBSCT eligible --Prior/Concurrent Therapy-- Biologic therapy: See Disease Characteristics No prior APBSCT with CD34 selected stem cells Chemotherapy: Not specified Endocrine therapy: Steroids must be discontinued at least 4 weeks prior to vaccination No concurrent steroids Radiotherapy: Not specified Surgery: Not specified Other: Any prior therapy must be completed at least 8 weeks prior to second APBSCT Recovered from the toxic effects of prior therapy No concurrent aspirin or nonsteroidal antiinflammatory drugs --Patient Characteristics-- Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: More than 8 weeks Hepatic: Bilirubin less than 2.0 mg/dL and not rising for at least 2-4 weeks before transplantation SGOT no greater than 4 times upper limit of normal and not rising for at least 2-4 weeks before transplantation Renal: Creatinine less than 2 times normal and not rising for at least 2-4 weeks before transplantation OR Creatinine clearance greater than 40 mL/min Cardiovascular: LVEF greater than 50% by MUGA scan Pulmonary: DLCO greater than 50% predicted Other: No other medical condition that would increase risk of transplantation HIV negative Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 1995-07; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry W. Kwak, Study Chair — National Cancer Institute (NCI)
Locations (3):
- United States (3):
  - Arkansas Cancer Research Center, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Medicine Branch, Bethesda, Maryland